CLINICAL TRIAL: NCT03101332
Title: Virtual Reality for Panic Disorder With Agoraphobia: a Clinical Trial
Brief Title: Virtual Reality for Panic Disorder With Agoraphobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR for panic with agoraphobia
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Panic; Agoraphobia
MeSH Terms: conditions — Agoraphobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-CBT (Experimental): Virtual Reality cognitive behavior therapy. 10-12 sessions of individual Cognitive Behavior Therapy with exposure tasks carried out through Virtual Reality.
  Interventions: Behavioral: Virtual Reality cognitive behavior therapy

INTERVENTIONS:
Behavioral: Virtual Reality cognitive behavior therapy — Cognitive interventions targeted to change catastrophic misinterpretations of the physiological symptoms that occur during a panic attack.
  Exposure via Virtual Reality to filmed sequences of environments typically feared by agoraphobic patients such as underground station/train, a tunnel, a lift and a public square, as well as exposure to the feared symptoms that occur in a typical panic attack.
  Interventions are delivered by a psychologist in face-to-face sessions.

SUMMARY:
Panic disorder with agoraphobia (PDA) is associated with considerable personal distress, functional disability and societal costs. A large number of studies have shown that Cognitive Behavior Therapy (CBT) is a highly effective treatment for PDA. However, the CBT-protocols proven to be most effective involves repeated exposure to the particular environments the agoraphobic patient fears such as trains, tunnels, lifts and shops. This cause great practical problems for health care services as such therapeutic efforts involves spending considerable time outside the clinic. For primary care services this is particularly challenging due to the large number of patients expected to be seen. Normally clinicians meet up to 7 patients daily which makes it almost practically impossible to offer 2-hour sessions, which is necessary to carry out the relevant exposure tasks. Hence, the treatment proven to be most effective, which primary care services are commissioned to deliver, is too comprehensive and time consuming to be applied in real practice.

The investigators believe that a possible solution to the above problem is to provide evidence-based CBT but with the exposure components carried out through Virtual Reality (VR) rather than in vivo. Some research has already been done with virtual reality and exposure therapy for anxiety disorders with promising results. The aim of this pilot study is to treat patients with agoraphobia with or with a history of panic disorder with a standardized exposure-based CBT-protocol through VR. The virtual environments that are used for the study are live sequences filmed in 360°. The investigators hypothesize that CBT with VR will be effective and lead to improvements on measures of panic disorder and agoraphobia.

ELIGIBILITY:
Inclusion:

* A primary diagnosis of Agoraphobia with or with a history of panic disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5).
* Minimum 18 years of age.
* Able to read and write in Swedish

Exclusion:

* Other primary axis-I disorder
* Ongoing substance abuse or addiction
* Current or previous episode of psychosis or bipolar disorder
* Severe major depressive disorder:
* Moderate to severe suicidal risk
* Non-stable antidepressant medication (changed during the last month) or not agreeing to keep dosage constant throughout the study
* Ongoing concurrent psychological treatment
* Having received previous high quality Cognitive Therapy or Cognitive Behavior Therapy for agoraphobia during the recent year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Mobility Inventory | Baseline, post-treatment (10 weeks), 6-month follow-up, 12-month follow-up
  Change at post-treatment (10 weeks), 6-month follow-up, and 12 month follow-up compared to baseline

SECONDARY OUTCOMES:
Panic disorder severity scale | Baseline, post-treatment (10 weeks), 6-month follow-up, 12-month follow-up
  Change at post-treatment (10 weeks), 6-month follow-up, and 12 month follow-up compared to baseline
Patient Health Questionnaire | Baseline, post-treatment (10 weeks), 6-month follow-up, 12-month follow-up
  Change at post-treatment (10 weeks), 6-month follow-up, and 12 month follow-up compared to baseline
World Health Organisation Disability Assessment Schedule | Baseline, post-treatment (10 weeks), 6-month follow-up, 12-month follow-up
  Change at post-treatment (10 weeks), 6-month follow-up, and 12 month follow-up compared to baseline
The World Health Organisation Quality of Life | Baseline, post-treatment (10 weeks), 6-month follow-up, 12-month follow-up
  Change at post-treatment (10 weeks), 6-month follow-up, and 12 month follow-up compared to baseline

OTHER OUTCOMES:
Presence Questionnaire | Week 1, week, 2, week3, week 4, week 5, week 6, week 7, week 8, week 9, week 10
  Means and standard deviations will be presented. No change is hypothesized for this measure

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Gustavsberg primary care center, Gustavsberg, Stockholm County
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No